CLINICAL TRIAL: NCT04732104
Title: Efficacy of Lidocaine and Xylometazoline Intranasal Spray in Anesthetizing Maxillary Teeth: An Open Label Randomized Controlled Trial
Brief Title: Efficacy of Lidocaine and Xylometazoline Intranasal Spray in Anesthetizing Maxillary Teeth
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Umair Wahid, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UWahid
Record Dates: First submitted 2021-01-14; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Effect of Drug
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intranasal spray anesthesia (Experimental): intranasal lidocaine lidocaine 4% topical
  Interventions: Drug: Lidocaine topical
- injectable local anesthesia (Active Comparator): gold standard infiltration local anesthesia (2% lidocaine with 1:100,000 epinephrine)
  Interventions: Drug: Lidocaine Hydrochloride

INTERVENTIONS:
Drug: Lidocaine topical — intranasal spray anesthesia will be administered for achieving pulpal local anesthesia of maxillary anterior and premolar teeth. Xylometazoline OTC decongestant will be used to prolong the duration of anesthesia
  Other Names: xylometazoline intranasal OTC decongestant
  Arms: intranasal spray anesthesia
Drug: Lidocaine Hydrochloride — injectable local anesthesia will be administered to achieve pulpal local anesthesia of maxillary anterior and premolar teeth
  Other Names: gold standard local anesthesia
  Arms: injectable local anesthesia

SUMMARY:
Different anesthetic techniques are used for achieving pulpal anesthesia of maxillary teeth. Recently tetracaine and oxymetazoline were used as local anesthetic agents in the form of an intranasal spray to achieve pulpal anesthesia of maxillary teeth. However tetracaine has its share of demerits, therefore we in our study have used lidocaine with xylometazoline in the form of an intranasal spray to achieve local anesthesia of maxillary anterior and premolar teeth for restorative procedures.

The objective of the study was to evaluate the efficacy of 4% lidocaine and 0.1% xylometazoline intranasal spray solution as compared to injectable 2% lidocaine with 1:100,000 epinephrine solution in anesthetizing maxillary anterior & premolar teeth for dental restorative procedures.

METHODS:

A total of 60 patients were enrolled in the study. Consecutive sampling was done for the study participants who met the inclusion criteria. 30 patients were randomized each to lidocaine/Xylometazoline or control local anesthesia group. Group A participants received 4% Lidocaine and 0.1% Xylometazoline solution as intranasal spray while Group B participants received injectable local anesthesia. Group 'A' participants received two doses of intranasal spray anesthesia four minutes apart. Local anesthesia was then assessed by probing soft tissues adjacent to the tooth and reading was taken on the Visual Analog Scale. If the reading was '0' the cavity preparation was performed. If the VAS reading was more than '0' a third dose of intranasal spray anesthesia was delivered. Local anesthesia was again assessed after ten minutes. If profound local anesthesia was still not achieved the case was labeled as failure of intranasal spray anesthesia and local anesthesia was achieved by conventional infiltration anesthesia. For Group B participants, local anesthesia was achieved by means of conventional infiltration anesthesia. Data were recorded on a designed proforma.

Chi-square test and Fischer exact test were applied to see the difference of efficacy among the two groups and any influence of variables (age group, gender, tooth location, cavity classification, ICDAS score or the number of sprays required to produce local anesthesia) on the efficacy.

DETAILED DESCRIPTION:
Different anesthetic techniques are used for achieving pulpal anesthesia of maxillary teeth. The most commonly used technique is the infiltration anesthesia that currently is the gold standard. However, infiltration uses a dental needle that is associated with its de merits also. This led to the discovery of novel methods to anesthetize teeth with smaller diameter needles or computerized delivery of local anesthesia. Recently tetracaine and oxymetazoline were used as local anesthetic agents in the form of an intranasal spray to achieve pulpal anesthesia of maxillary teeth. However tetracaine has its share of demerits, therefore we in our study have used lidocaine with xylometazoline in the form of an intranasal spray to achieve local anesthesia of maxillary anterior and premolar teeth for restorative procedures.

OBJECTIVES:

The objective of the study was to evaluate the efficacy of 4% lidocaine and 0.1% xylometazoline intranasal spray solution as compared to injectable 2% lidocaine with 1:100,000 epinephrine solution in anesthetizing maxillary anterior & premolar teeth for dental restorative procedures.

METHODS:

This open label randomized controlled trial was performed at the Department of Operative Dentistry, Dr.Ishrat Ul Ebad Khan Institute of Oral Health Sciences, Dow University of Health Sciences Karachi between July 2018 and June 2020.

A total of 60 patients were enrolled in the study. Consecutive sampling was done for the study participants who met the inclusion criteria. 30 patients were randomized each to lidocaine/Xylometazoline or control local anesthesia group. Group A participants received 4% Lidocaine and 0.1% Xylometazoline solution as intranasal spray while Group B participants received injectable local anesthesia. Group 'A' participants received two doses of intranasal spray anesthesia four minutes apart. Local anesthesia was then assessed by probing soft tissues adjacent to the tooth and reading was taken on the Visual Analog Scale. If the reading was '0' the cavity preparation was performed. If the VAS reading was more than '0' a third dose of intranasal spray anesthesia was delivered. Local anesthesia was again assessed after ten minutes. If profound local anesthesia was still not achieved the case was labeled as failure of intranasal spray anesthesia and local anesthesia was achieved by conventional infiltration anesthesia. For Group B participants, local anesthesia was achieved by means of conventional infiltration anesthesia. Data were recorded on a designed proforma.

SPSS v16 was used to analyze the data with level of significance set at p<0.05. Demographic data were analyzed upon the basis of frequency and percentages. Chi-square test and Fischer exact test were applied to see the difference of efficacy among the two groups and any influence of variables (age group, gender, tooth location, cavity classification, ICDAS score or the number of sprays required to produce local anesthesia) on the efficacy.

ELIGIBILITY:
INCLUSION CRITERIA

* Adults aged 18-40 years,
* Patients having a vital maxillary premolar, canine or incisor.
* Patients having Class 1,2,3,4 or 5 restorations (G.V. Black).95
* Patients having heart rate between 55 and 100 beats per min.
* Patients with a seated Systolic blood pressure between 95 and 150 mm Hg and diastolic blood pressure between 60 and 100 mm of Hg. (Although short-term use of topical alpha-2 agonists like xylometazoline has no systemic toxicity and are available as over the counter drugs but long-term abuse has been reported to cause systemic vasoconstriction and cardiovascular complications like hypertensive crisis therefore the cut off limit has been selected for blood pressure).
* Teeth with no radiographic evidence of pulpal or periapical pathosis.
* Patients having ICDAS caries detection score of 4, 5 or 6.
* Patients who fulfilled alcohol sniff test criterion.

EXCLUSION CRITERIA

* Patients with Upper respiratory tract infection.
* Patients with Uncontrolled thyroid disease.
* Patients having a known allergy to any of the components used in the solution.
* Pregnant or breast feeding patients.
* Those patients having 5 or more nosebleeds per month.
* Patients who received any local anesthetic/analgesic within 24 hours of study drug administration.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Achievement of local anesthesia | First reading on VAS will be taken after administering 2 intranasal sprays i.e. 14 minutes after administration of the first spray
  local anesthesia will be assessed with the help of Visual Analog Scale. VAS score must be '0' before cavity preparation must begin
Achievement of local anesthesia | If needed, second reading on VAS will be taken after administering 3 intranasal sprays i.e. 24 minutes after administration of the first spray
  local anesthesia will be assessed with the help of Visual Analog Scale. VAS score must be '0' before cavity preparation must begin

CONTACTS AND LOCATIONS:
Overall Officials: Umair Wahid, MDS, Principal Investigator — DUHS
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT04732104/Prot_SAP_ICF_000.pdf